CLINICAL TRIAL: NCT01472224
Title: Volume Measurement and Progression Surveillance of Intracerebral Haemorrhage Using Transcranial Ultrasound
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Hanne Christensen, Associate Research Professor, Consultant neurologist, Bispebjerg Hospital
Other Study IDs: H-1-2011-069
Record Dates: First submitted 2011-11-13; First posted 2011-11-16 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Stroke; Cerebral Hemorrhage
Keywords: Transcranial ultrasound; Haematoma expansion
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study investigates the ability of ultrasound to measure the volume of a brain hemorrhage in the acute phase after hospital admission.

It is known that approximately 30% of patients admitted with a brain hemorrhage will suffer from enlargement of the hematoma within the first hours after admission.

In this study the investigators measure the volume of the hematoma every 30 minutes up to 6 hours after admission and every 2 hours between 6-12 hours.

DETAILED DESCRIPTION:
This study investigates the use of transcranial ultrasound (TCU) for the surveillance of patients with intracerebral hemorrhages. Using transcranial ultrasound makes it possible to visualize and follow the bleeding progression through 3 points of the scull where the bone is thin enough to allow the penetration of sound waves. This can be done at bedside. Today the investigators do not know for sure if clinical parameters determine a haematoma expansion. TCU will allow us to follow the haematoma progression serially in the acute phase and relate the haematoma expansion to parameters like blood pressure, neurological status (NIHSS-score) and radiological signs of ongoing bleeding (spot signs) on CT-angiogram (CTA).

Hypothesis:

1. Bedside ultrasound volume assessment is accurate in estimating the haematoma volume compared to computer tomography (CT) and can dynamically document the haematoma expansion.
2. The haematoma expansion is accompanied by neurological deterioration and happens only with patients with CT demonstrated spot signs.
3. The haematoma expansion is observed with patients with high blood pressure.

Aim of study:

1. To validate the accuracy of ultrasound (US) compared to CT in estimating haematoma volume with ICH patients.
2. To measure ICH volume serially in the acute phase using US and up to 12 hours aiming at:

   * Describing the timing of the haematoma expansion.
   * Relating to neurological deterioration, systemic blood pressure and detection of spot signs on CTA.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Bispebjerg Hospital stroke unit with CT demonstrated spontaneous ICH
* Hospital admission within 4,5 hours after symptom onset
* CTA on admission
* GCS>8 (non-comatose)

Exclusion Criteria:

* Lack of informed consent
* Underlying Pathology (tumor, AVM, aneurism)
* Lack of temporal bone window

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely admitted stroke patients with intracerebral hemorrhage. Hemorrhage not older than 4,5 hours
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Christensen, MD, Ph.D, DMSci, Principal Investigator — Bispebjerg Hospital - Department of neurology
Locations (1):
- Bispebjerg Hospital, Neurologisk afdeling, Copenhagen, Region H, Denmark

REFERENCES:
- [Background] Mayer SA, Rincon F. Treatment of intracerebral haemorrhage. Lancet Neurol. 2005 Oct;4(10):662-72. doi: 10.1016/S1474-4422(05)70195-2. PMID 16168935
- [Background] Brott T, Broderick J, Kothari R, Barsan W, Tomsick T, Sauerbeck L, Spilker J, Duldner J, Khoury J. Early hemorrhage growth in patients with intracerebral hemorrhage. Stroke. 1997 Jan;28(1):1-5. doi: 10.1161/01.str.28.1.1. PMID 8996478
- [Background] Broderick JP, Brott TG, Duldner JE, Tomsick T, Huster G. Volume of intracerebral hemorrhage. A powerful and easy-to-use predictor of 30-day mortality. Stroke. 1993 Jul;24(7):987-93. doi: 10.1161/01.str.24.7.987. PMID 8322400
- [Background] Davis SM, Broderick J, Hennerici M, Brun NC, Diringer MN, Mayer SA, Begtrup K, Steiner T; Recombinant Activated Factor VII Intracerebral Hemorrhage Trial Investigators. Hematoma growth is a determinant of mortality and poor outcome after intracerebral hemorrhage. Neurology. 2006 Apr 25;66(8):1175-81. doi: 10.1212/01.wnl.0000208408.98482.99. PMID 16636233
- [Background] Leira R, Davalos A, Silva Y, Gil-Peralta A, Tejada J, Garcia M, Castillo J; Stroke Project, Cerebrovascular Diseases Group of the Spanish Neurological Society. Early neurologic deterioration in intracerebral hemorrhage: predictors and associated factors. Neurology. 2004 Aug 10;63(3):461-7. doi: 10.1212/01.wnl.0000133204.81153.ac. PMID 15304576
- [Background] Ohwaki K, Yano E, Nagashima H, Hirata M, Nakagomi T, Tamura A. Blood pressure management in acute intracerebral hemorrhage: relationship between elevated blood pressure and hematoma enlargement. Stroke. 2004 Jun;35(6):1364-7. doi: 10.1161/01.STR.0000128795.38283.4b. Epub 2004 Apr 29. PMID 15118169
- [Background] Kothari RU, Brott T, Broderick JP, Barsan WG, Sauerbeck LR, Zuccarello M, Khoury J. The ABCs of measuring intracerebral hemorrhage volumes. Stroke. 1996 Aug;27(8):1304-5. doi: 10.1161/01.str.27.8.1304. PMID 8711791
- [Background] Thompson AL, Kosior JC, Gladstone DJ, Hopyan JJ, Symons SP, Romero F, Dzialowski I, Roy J, Demchuk AM, Aviv RI; PREDICTS/Sunnybrook ICH CTA Study Group. Defining the CT angiography 'spot sign' in primary intracerebral hemorrhage. Can J Neurol Sci. 2009 Jul;36(4):456-61. doi: 10.1017/s0317167100007782. PMID 19650356
- [Background] Becker G, Winkler J, Hofmann E, Bogdahn U. Differentiation between ischemic and hemorrhagic stroke by transcranial color-coded real-time sonography. J Neuroimaging. 1993 Jan;3(1):41-7. doi: 10.1111/jon19933141. PMID 10148076
- [Background] Kern R, Kablau M, Sallustio F, Fatar M, Stroick M, Hennerici MG, Meairs S. Improved detection of intracerebral hemorrhage with transcranial ultrasound perfusion imaging. Cerebrovasc Dis. 2008;26(3):277-83. doi: 10.1159/000147456. Epub 2008 Jul 23. PMID 18648201
- [Background] Maurer M, Shambal S, Berg D, Woydt M, Hofmann E, Georgiadis D, Lindner A, Becker G. Differentiation between intracerebral hemorrhage and ischemic stroke by transcranial color-coded duplex-sonography. Stroke. 1998 Dec;29(12):2563-7. doi: 10.1161/01.str.29.12.2563. PMID 9836768
- [Background] Perez ES, Delgado-Mederos R, Rubiera M, Delgado P, Ribo M, Maisterra O, Ortega G, Alvarez-Sabin J, Molina CA. Transcranial duplex sonography for monitoring hyperacute intracerebral hemorrhage. Stroke. 2009 Mar;40(3):987-90. doi: 10.1161/STROKEAHA.108.524249. Epub 2009 Jan 22. PMID 19164795
- [Background] Seidel G, Kaps M, Dorndorf W. Transcranial color-coded duplex sonography of intracerebral hematomas in adults. Stroke. 1993 Oct;24(10):1519-27. doi: 10.1161/01.str.24.10.1519. PMID 8378956
- [Derived] Ovesen C, Christensen AF, Krieger DW, Rosenbaum S, Havsteen I, Christensen H. Time course of early postadmission hematoma expansion in spontaneous intracerebral hemorrhage. Stroke. 2014 Apr;45(4):994-9. doi: 10.1161/STROKEAHA.113.003608. Epub 2014 Mar 13. PMID 24627116